CLINICAL TRIAL: NCT06294171
Title: Efficacy of Modified Piezosurgery Alveolar Bone Cut With Osseodensification Drills in Expanding Narrow Alveolar Bone (Randomized Clinical Trial)
Brief Title: Efficacy of Modified Piezosurgery Alveolar Bone Cut With Osseodensification Drills in Expanding Narrow Alveolar Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Amjed Kadhim Tayyeh, Bachelor's dental Surgery ( B. D. S), University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Modified Alveolar Bone Cut
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Dental Implant Failed
Keywords: peizosurgery , osseodensification , modified ridge splitting , dental implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- measurement of alveolar ridge width (Other): the surgical procedure started with envelop flap reflection. A mucoperiosteal elevator was used to reflect the buccal and palatal flaps that were enough to expose the crestal part of alveolar ridge with clear visibility and accessibility. Measuring the width of the alveolar ridge 1 mm below the crest using bone caliber. Using piezoelectric surgery unit (Piezosurgery Ultrasonic® mectron, Italy), a horizontal crestal cut was produced along the crest of the bone. The cut depth extended into the same depth of the final dental implant to be inserted and then Versah Drills will be used in a successive manner and under copious irrigation with chilled sterile normal saline.We will measure the rate of ridge expansion by bone caliber to determine the efficacy of combining Versah drills with piezo surgery in expanding narrow alveolar bone.
  Interventions: Device: measurement of alveolar ridge width

INTERVENTIONS:
Device: measurement of alveolar ridge width — the surgical procedure started with envelop flap reflection. A mucoperiosteal elevator was used to reflect the buccal and palatal flaps that were enough to expose the crestal part of alveolar ridge with clear visibility and accessibility. Measuring the width of the alveolar ridge 1 mm below the crest using bone caliber. Using piezoelectric surgery unit (Piezosurgery Ultrasonic® mectron, Italy), a horizontal crestal cut was produced along the crest of the bone. The cut depth extended into the same depth of the final dental implant to be inserted and then Versah Drills will be used in a successive manner and under copious irrigation with chilled sterile normal saline.We will measure the rate of ridge expansion by bone caliber to determine the efficacy of combining Versah drills with piezo surgery in expanding narrow alveolar bone.

SUMMARY:
The aim of the study is to determine the efficacy of modified piezosurgery with osseodensification drills in expanding narrow alveolar bone.

DETAILED DESCRIPTION:
Atrophic maxilla or mandible can lead to lack of prosthesis retention because of an inadequate bearing area causing both functional and physiological problems for patient, these problems can be treated for patient satisfaction with an implant supported fixed or removable complete or partial denture. Atrophic edentulous jaws can represent a significant challenge to the successful use of endosseous implants for prosthetic reconstruction of the edentulous mandible.

A collapsed alveolar ridge demonstrating a narrow width (less than 5 mm in many cases) and grossly adequate alveolar height is the most common candidate for the RSP.

Beginners in RSP should initially choose a 4-5 mm thickness of an even maxillary alveolar ridge and strive to almost double it in width.

A 3-mm alveolar ridge generally consists of 3 thin bone layers (in a horizontal sandwich fashion): 2 cortical plates (about 1 mm each) separated by 1 cancellous layer (about 1 mm). The wider the cancellous bone layer (the layer where the split is done), the easier it will be to accomplish the RSP

ELIGIBILITY:
Inclusion criteria:

1. Patient's age ≥18 years.
2. Absence of any medical disease that compromise wound healing.
3. Patient with good oral hygiene.
4. Narrow alveolar bone (3-4 mm) with minimum alveolar bone height of (12 mm).

Exclusion criteria:

1. Uncontrolled medically compromised patients.
2. Heavy smokers (> 10 cigarettes per day).
3. Patient with parafunctional habits.
4. Local infection at implant site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
expansion rate | immediately
  by digital vernier
expansion rate | after 6 months
  by digital vernier

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
It will be mostly available on request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 11/11/2024 for 3 month
Access Criteria: I can provide data as word